CLINICAL TRIAL: NCT01255267
Title: The Correlation Between Genetic Polymorphism, Platelet Activity, , Clopidogrel Responsiveness, and Serum Adipokine Concentration in Asian Acute Coronary Syndrome Patients
Brief Title: The Correlation Between Genetic Polymorphism, Platelet Activity, Clopidogrel Responsiveness, and Serum Adipokine Concentration in Asian Acute Coronary Syndrome Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Other Study IDs: DMR99-IRB-041
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Acute Coronary Syndrome; Chronic Coronary Artery Disease
Keywords: Acute coronary syndrome and chronic coronary artery disease patients
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Acute coronary syndrome patients
- Chronic coronary artery disease patients
- Healthy control

SUMMARY:
In this study, we evaluate the acute coronary syndrome patients to see if there is correlation between platelet activity, genetic polymorphism (CYP2C19 and ABCB1), serum adipokines level, and Clopidogrel responsiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 y/o
2. Acute coronary syndrome patients
3. Chronic coronary artery disease patients
4. Healthy volunteers

Exclusion Criteria:

1. Patient refusal
2. Allergy to Clopidogrel
3. Receive Gp IIb/IIIa inhibitor simultaneously
4. Cancer history
5. Severe renal and liver function impairment
6. Coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute coronary syndrome and chronic coronary artery diseae patients
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan